CLINICAL TRIAL: NCT00622401
Title: Vaccination of Patients With Breast Cancer With Dendritic Cell/Tumor Fusions and IL-12
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: Dana-Farber Cancer Institute (Other); Brigham and Women's Hospital (Other); Harvard Medical School (HMS and HSDM) (Other); United States Department of Defense (U.S. Federal Agency); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Avigan, MD, Principal Investigator, Dana-Farber Cancer Institute
Organization: Dana-Farber Cancer Institute (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-221; NCI 6040; U01CA062490 (NIH); P30CA006516 (NIH); NCT00731406 (obsolete NCT alias)
Record Dates: First submitted 2008-02-14; First posted 2008-02-25 (Estimated); Results first posted 2016-03-16 (Estimated); Last update posted 2017-11-14 (Actual); Status verified 2017-10

CONDITIONS: Breast Cancer
Keywords: stage IV breast cancer; dendritic cell vaccine; tumor fusion vaccine; IL-12
MeSH Terms: conditions — Breast Neoplasms | interventions — Interleukin-12

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group 1 (Experimental): Dendritic Cell/Tumor Fusion Vaccine Only
  Interventions: Biological: Dendritic Cell/Tumor Fusion Vaccine
- Group 2 (Experimental): Dendritic Cell/tumor fusion vaccine and low dose IL-12
  Interventions: Biological: Dendritic Cell/Tumor Fusion Vaccine; Drug: Interleukin-12
- Group 3 (Experimental): Dendritic Cell/tumor fusion vaccine and higher dose IL-12
  Interventions: Biological: Dendritic Cell/Tumor Fusion Vaccine; Drug: Interleukin-12

INTERVENTIONS:
Biological: Dendritic Cell/Tumor Fusion Vaccine — Vaccine is derived from the participants dendritic cells and tumor cells
  Other Names: DC/tumor cell fusion vaccine
Drug: Interleukin-12 — Given subcutaneously at dose of 30ng/kg
  Other Names: IL-12; rhIL-12
  Arms: Group 2
Drug: Interleukin-12 — Given subcutaneously at dose of 100ng/kg
  Other Names: IL-12; rhIL-12
  Arms: Group 3

SUMMARY:
The purpose of this study is to test the safety of an investigational Dendritic Cell/Tumor Fusion vaccine given with IL-12 for patients with breast cancer.

RATIONALE: Vaccines made from a person's tumor cells and white blood cells may help the body build an effective immune response to kill tumor cells. Interleukin-12 may stimulate the white blood cells to kill tumor cells. Giving vaccine therapy together with interleukin-12 may kill more tumor cells.

PURPOSE: This phase I/II trial is studying the side effects and best dose of interleukin-12 when given together with vaccine therapy and to see how well they work in treating women with stage IV breast cancer.

DETAILED DESCRIPTION:
TUMOR COLLECTION: Tumor cells will be collected from the participant to make the study vaccine. Based on the location of the tumor, a decision will be made as to the best approach to obtain these cells.

DENDRITIC CELL COLLECTION: Participants will undergo a procedure known as leukapheresis to obtain their dendritic cells (this procedure may be done before or after the tumor cells have been obtained). This procedure takes about 2-4 hours. If not enough cells are collected, the participant may be asked to return for an additional leukapheresis procedure. If sufficient number of cells are obtained, tumor cells and dendritic cells will then be fused (combined together to make one larger cell) together in the laboratory and divided into the appropriate dose for administration.

TREATMENT: Treatment will consist of an injection of tumor cells fused with dendritic cells under the skin every 3 weeks for a total of 9 weeks. The dose that the participant receives will depend on the total number of fusion cells that are made.

STUDY COHORTS: The first group of three participants will receive the DC/Tumor Fusion study vaccine alone. The next group of 3 participants will receive the DC/Tumor Fusion study vaccine with a low dose of Il-12. If there are no significant side effects the following groups of subjects will be treated with the DC/Tumor Fusion study vaccine and a higher dose of Il-12.

PATIENT MONITORING: Participants will be carefully monitored during the study period and the following tests and procedures will be performed: physical exams (weekly); blood collections (weekly); DC/Tumor Fusion study vaccine Journal (for the participant to record any side effects or other medications they may be taking); tumor cells skin test (before the first vaccine and one month following the last vaccine); skin biopsy at the site of the vaccination administration, accessible tumor site, or if there is a local reaction site.

ELIGIBILITY:
Inclusion Criteria:

* Stage IV breast cancer with measurable disease and accessible tumor
* ECOG Performance Status 0-2 with greater than six week life expectancy
* 18 years of age or older
* Laboratory values as outlined in the protocol

Exclusion Criteria:

* Patients must not have received other immunotherapy treatment in the three months prior to the initial vaccination
* Patients may not be on herceptin therapy during this protocol and may not have received it for four weeks prior to initial vaccination
* Patients must not have received weekly chemotherapy or hormonal treatment for two weeks prior to the initial vaccination and must not have received monthly chemotherapy for four weeks prior to the initial vaccination
* Clinical evidence of CNS disease
* Clinically significant autoimmune disease
* Patients who are HIV+
* Serious intercurrent illness such as infection requiring IV antibiotics, or significant cardiac disease characterized by significant arrhythmia, ischemic coronary disease or congestive heart failure
* Pregnant of lactating women will be excluded, all premenopausal women must undergo pregnancy testing

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-12; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Avigan, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: Dendritic Cell/Tumor Fusion Vaccine Only: Dendritic Cell/Tumor Fusion Vaccine Only
  Dendritic Cell/Tumor Fusion Vaccine: Vaccine is derived from the participants dendritic cells and tumor cells
- Group 2: Dendritic Cell/Tumor Fusion Vaccine and Low Dose IL-1: Dendritic Cell/tumor fusion vaccine and low dose IL-12
  Dendritic Cell/Tumor Fusion Vaccine: Vaccine is derived from the participants dendritic cells and tumor cells
  Interleukin-12: Given subcutaneously at dose of 30ng/kg
- Group 3: Dendritic Cell/Tumor Fusion Vaccine and Higher Dose I: Dendritic Cell/tumor fusion vaccine and higher dose IL-12
  Dendritic Cell/Tumor Fusion Vaccine: Vaccine is derived from the participants dendritic cells and tumor cells
  Interleukin-12: Given subcutaneously at dose of 100ng/kg
Period: Overall Study
Arm/Group | Group 1: Dendritic Cell/Tumor Fusion Vaccine Only | Group 2: Dendritic Cell/Tumor Fusion Vaccine and Low Dose IL-1 | Group 3: Dendritic Cell/Tumor Fusion Vaccine and Higher Dose I
Started | 6 | 2 | 0 (Never Opened)
Completed | 3 | 0 | 0
Not Completed | 3 | 2 | 0
Not completed — Disease progression prior to treatment | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Population: Females >18yo with metastatic breast cancer
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: Dendritic Cell/Tumor Fusion Vaccine Only | Group 2: Dendritic Cell/Tumor Fusion Vaccine and Low Dose IL-1 | Group 3: Dendritic Cell/Tumor Fusion Vaccine and Higher Dose I | Total
Number analyzed (Participants) | 6 | 2 | 0 | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 |  | 0
  Between 18 and 65 years | 4 | 2 |  | 6
  >=65 years | 2 | 0 |  | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 2 |  | 8
  Male | 0 | 0 |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 2 |  | 8

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events Associated With Vaccination of Breast Cancer Patients With Dendritic Cell (DC)/Tumor Fusion Vaccine
Description: Using CTCAE version 3, adverse events associated with the intervention were captured throughout the treatment portion of the study. All adverse events were then compiled and the number of patients who experienced these adverse events was recorded.
Time Frame: 3 years
Population: All three patients experienced adverse events that were determined to be at least possibly related to the vaccine. The number of times each toxicity was observed is captured in the adverse events section.
Measure: Number; unit: participants
Arm/Group | Group 1
Number analyzed (Participants) | 3
participants | 3

2. Secondary Outcome: To Determine if Cellular and Humoral Immunity is Induced by Serial Vaccination With DC/Tumor Fusion Cells and rhIL-12.
Description: This outcome was not measured because no patients were treated with rhIL-12.
Time Frame: 3 years
Population: This outcome was not measured because no patients were treated with rhIL-12.
Arm/Group | Group 1: Dendritic Cell/Tumor Fusion Vaccine Only | Group 2: Dendritic Cell/Tumor Fusion Vaccine and Low Dose IL-1 | Group 3: Dendritic Cell/Tumor Fusion Vaccine and Higher Dose I
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Group 1
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 3/3
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=3)
Vaccine Site Reaction (Investigations) | 2 (3)
Nausea (Gastrointestinal disorders) | 1 (2)
Myalgias (General disorders) | 1 (1)
Rash (General disorders) | 1 (1)
Pain (Nervous system disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
In the conduct of the study, it became apparent that the setting of advanced breast cancer with malignant effusions/ascites for vaccine generation was a difficult setting for evaluation of an immune based therapy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No